CLINICAL TRIAL: NCT01500967
Title: Shi-style Cervical Manipulations for Cervical Radiculopathy-A Randomized Single Blinded Controlled Trial
Brief Title: Shi-style Cervical Manipulations for Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Cui xuejun, Longhua Hospital, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Manual Therapy for Cervicalgia
Record Dates: First submitted 2011-08-30; First posted 2011-12-29 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traction (Active Comparator): 6kg to 10kg, 3 times a week, once the other day（except the weekends）,20 minutes, 2 weeks.
  Interventions: Other: Cervical Traction control
- Manipulations (Experimental): Shi-style manipulations is a cervical manipulation for cervical radiculopathy.This manipulation is a kind of traditional Chinese massage and it can dredge the meridians. Patients are treated every day for 30 minutes. Seven times as one course and totally there are two courses. 3 times a week, once the other day（except the weekends）,30 minutes, 2 weeks.
  Interventions: Other: Shi-style cervical manipulations

INTERVENTIONS:
Other: Shi-style cervical manipulations — Shi-style cervical manipulation is a spinal manipulation for cervical radiculopathy.It is a kind of traditional chinese massage and can dredge the meridian.Patients are treated every day for 30 minutes.Seven times at one course and totally there are two courses.3 times a week, once the other day（except the weekends）,30 minutes, 2 weeks.
  Other Names: manipulations for cervical radiculopathy
  Arms: Manipulations
Other: Cervical Traction control — 6kg to 10kg, 3 times a week, once the other day（except the weekends）,20 minutes, 2 weeks.
  Other Names: Cervical traction
  Arms: Traction

SUMMARY:
Neck pain and related problems occur frequently in modern societies and have a considerable impact on individuals and the society. Cervical radiculopathy (CR) generally presents with pain, numbness, or weakness in a dermatomal distribution. CR results from impingement on a nerve root by either spondylotic narrowing of the neural foramen or a lateral intervertebral disc herniation. Various studies have shown that nonoperative management for CR is effective, such as medications, physical therapy, Spinal manipulation, traction, acupuncture, collar immobilization and epidural steroid injections. Spinal manipulation is one of the manual techniques for treating mechanical neck pain. No high-quality evidence has proved the effectiveness of manipulative therapy in the treatment of cervical radiculopathy. However, limited evidence suggests that manipulation may provide short-term benefit in the treatment of neck pain, cervicogenic headaches and radicular symptoms. Few complications, such as worsening radiculopathy, myelopathy, and spinal cord injury, may occur. Spinal massage manipulation is used for centuries in China. Many patients with cervical disc disease are increasingly turning to manipulations to alleviate their symptoms and reduce the side effects of medications. The goal of this study is to determine the efficacy of a spinal manipulation, three steps and nine manipulations, on treating with the cervical radiculopathy.

DETAILED DESCRIPTION:
Radiculopathy generally presents with pain, numbness, or weakness in a dermatomal distribution. Causative factors include an acute nucleus pulposus herniation, spondylitic changes around the foramen causing nerve compression, or a combination of these.

Cervical radiculopathy results from impingement on a nerve root by either spondylotic narrowing of the neural foramen or a lateral intervertebral disc herniation. Frequent complaints include painful neck movements, radicular pain, paraspinal muscle spasm, muscle weakness, and diminished deep tendon reflexes (Radhakrishnan K, 1994). Radiculopathy tends to produce substantial limitation of movement of the head and neck.

The goals of any treatment plan should be well defined. Specifically, it should be the goal of the treating physician to relieve pain, improve function, and prevent recurrence. Although some symptomatic patients meet surgical criteria, most patients are clearly candidates for nonoperative treatment. Treatment modalities for radiculopathy include rest, medications, physical therapy, manipulation, injections, and patient education.

Various studies have shown that nonoperative management of cervical radiculopathy leaves a substantial minority of patients with persistently troublesome symptoms (Lees F, 1963,41, 42). Lees and Turner found that in two thirds of patients, symptoms tend to persist in the absence of surgical treatment (Lees F, 1963). DePalma and Subin found that of 255 patients treated nonoperatively, only 29% experienced complete symptom relief (Radhakrishnan K, 1994,41). Better outcomes with nonoperative management, however, have been observed in studies that were based in physiotherapy centers than those from surgical series (Radhakrishnan K, 1994).

Spinal balance is the way Professor Shi Qi " Arthralgia theory" and " The theory of muscle imbalance " theory under the guidance of mix martial arts, Wang Shi expertise and Traumatology, combined with clinical experience and experimental research. Rub, take, roll, put, loose, pull, friction, shaking, pinching, so called "nine manipulations." It can adjust qi and blood, phlegm stasis, Dredge meridians, spasm pain, support organs, alleviate, correct cervical dynamic and static imbalance. Three steps and nine manipulations is the common method of treatment of Professor Shi Qi for cervical disease .

ELIGIBILITY:
Inclusion Criteria:

* Informed consent and signed an informed consent;
* aged 18 to 65 year-old male or female ;
* appear cervical nerve root symptoms typical of 3 months to 5 years;
* VAS pain greater than 30 mm.
* positive for one of the following :Brachial plexus traction test, Foraminal compression test, Neck rotation test is less than 60 degrees, Foraminal separation test, Decreased muscle strength.

Exclusion Criteria:

* nerve root in the past received surgical treatment of cervical or neck trauma;
* with obvious symptoms of vertigo, TCD examination there was abnormal;
* signs and symptoms of spinal cord compression, MRI found that spinal cord oppressors[e];
* pregnant women, lactating women;
* can not attend follow-up (such as six months or less distance of immigrant relocation plan, no mobile phones and other communication tools, etc.), and no ability to participate in six months follow-up of patients;
* currently participating in cervical spondylosis associated with other clinical trials;
* hepatic, renal, hematopoietic system, endocrine system, cardiovascular, nervous system, primary and other serious diseases, tuberculosis, vertebral deformities, cancer and mental illness;
* There are opioid analgesics, sedative hypnotics and alcohol abuse history;
* those who can not read and write Chinese.
* the past two weeks received RF, minimally invasive , ozone , a small knife , or other manual therapy and Closed injection treatment.
* vertebral displacement, forward, backward or lateral horizontal displacement > 3 mm, the angulation between adjacent intervertebral > 11 °.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 648 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | changes from baseline at 2 weeks

SECONDARY OUTCOMES:
SF 36 | changes from baseline at 2 weeks
Visual Analogue Scale | changes from baseline at 2 weeks
Neck Disability Index | changes from baseline at 4 weeks
SF 36 | 4 weeks
Visual Analogue Scale | 4 weeks
Neck Disability Index | changes from baseline at 3 months
SF 36 | changes from baseline at 3 months
Visual Analogue Scale | changes from baseline at 3 months
Neck Disability Index | changes from baseline at 6 months
SF 36 | changes from baseline at 6 months
Visual Analogue Scale | changes from baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, MD, Principal Investigator — Shanghai University of Traditional Chinese Medicine
Locations (1):
- Longhua Hospital, Shanghai, Shanghai Municipality, China